CLINICAL TRIAL: NCT05088551
Title: The Effect of the Educational Plan Prepared According to the Health Literacy Levels of Patients With Total Knee Arthroplasty on the Healing Process and the Quality of Life: Randomized Controlled Study
Brief Title: The Effect of the Educational Plan Prepared According to the Health Literacy Levels of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Nilgun Ozbas, Assistant Professor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14574941- 199-27487
Record Dates: First submitted 2021-09-04; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Total Knee Arthroplasty; Patient Education
Keywords: Total knee arthroplasty; Patient education; Nursing; Health literacy; Quality of life
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants, care providers were left blind. At the same time in the statistical analysis and reporting phase, the researchers were left blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): When the patients were admitted to the clinic,and the face-to-face interview method and the Patient Information Form,Turkey Health Literacy Scale-32,Patient Learning Needs Scale,Functional Assessment Form and Quality of Life Scale Form were filled.The second interview was conducted on the second or third day after the surgery, just before the patients were discharged.The Functional Assessment Form,Discharge Data Collection Form, and Quality of Life Questionnaire were applied.The third interview was performed 15 days after the surgery when the patients came for control or by phone.The 15th Day Recovery Process Data Collection Form were applied.The last interview was carried out six weeks after the surgery,either face-to-face or by phone,and the Functional Assessment Form,6th Week Post-Discharge Recovery Process Data Collection Form,and Quality of Life Questionnaire were applied again.Except for the routine practices of the service,no intervention was made to the control group patients.
- Intervention group (Experimental): Unlike the control group, the intervention group was given the education plan prepared by the researcher after filling out the forms when the patients were first encountered, and the education was carried out using various training methods such as lecture, question-answer, demonstration, and practice.Patients whose check-up time after discharge was nearing (15 days after the operation) were called a few days before and their visit time was learned. The forms were filled in by interviewing the patients face-to-face by the researcher on the 15th day and the 6th week after the operation or making a phone call on the same day with the patients who could not be reached.
  Interventions: Other: Patient Education

INTERVENTIONS:
Other: Patient Education — The education was divided into three parts. The information in the first part of the booklet (general information, preoperative preparation, and operation day) is given in the preoperative period. In the postoperative period, the patients were visited and the information in the second part (postoperative hospital stay, first, second, and third-day goals after surgery) was given. Before the patients were discharged, the information in the third section (things to be considered in the recovery process at home) was presented. According to the physical conditions of the clinic, patient education was carried out in an area suitable for teaching as much as possible.
  Arms: Intervention group

SUMMARY:
The reasons such as the advanced age of most patients with Total Knee Arthroplasty (TKA), the presence of concomitant diseases, and bilateral prostheses cause a decrease in the quality of life by negatively affecting the healing processes of the patients. Patients who try to adapt to the problems experienced during postoperative recovery need the information to develop coping behaviors. Nurses play a crucial role in ensuring adequate and effective access of information to the patient during this challenging process, which significantly affects mobility and, consequently, life activities. Effective educational interventions to be implemented by nurses enable patients to make decisions about health problems and act to improve their quality of life. However, for patient education to be efficient, the information given must be easy to read, understandable, and suitable for various learning styles to cope with problems more effectively. Still, individuals with low health literacy have problems benefiting from all services provided, exceptionally patient education, at the desired level.

DETAILED DESCRIPTION:
Patients with TKA face many problems in the early postoperative period and home processes after discharge. In this process, the instruction that will be given by nurses as a part of the care is critical. Patient education will contribute to less stress for patients, effective participation in their care, and more minor problems in the recovery process at home after discharge and increase positive patient outcomes. However, for the teaching to be effective, nurses must first determine the health literacy levels of individuals. When initiatives are planned following the level of health literacy, it is thought that individuals' adaptation to the duration of their health will increase, the process will progress effectively, the recovery will be positively affected, and the quality of life will increase. Accordingly, this study was conducted to examine the effect of the curriculum prepared according to patients' health literacy levels with TKA on the healing process and quality of life.

Research hypotheses:

H1a- Patient education, which is planned according to health literacy levels, positively affects patients' quality of life.

H1b- Patient education, which is planned according to health literacy levels, reduces patients' problems on the 15th day after surgery.

H1c- Patient education, which is planned according to health literacy levels, reduces patients' problems in the 6th week after surgery.

H1d- Patient education, which is planned according to health literacy levels, affects the postoperative improvement in functional status in patients.

Study Design: A control group intervention research. Method: 102 patients, 51 experimental groups, and 51 control groups participated in the study. The sample was chosen randomly from the universe by the researcher. From the patients hospitalized in the clinic and matching the research criteria, the control group was determined by random method according to the order of the patients, and their data were collected. Then, the intervention group data were obtained, paying attention to the similarity of the groups in terms of education, age, and gender. In the study, the education plan prepared in line with the control group data was applied to the intervention group, and its effects on the healing processes were observed.

Data were collected with Patient Introduction, Patient Learning Requirements, Functional Evaluation, Turkey Health Literacy, Discharge Data Collection, Post-Discharge 15th and Sixth Week Recovery Process Data Collection, Quality of Life Forms.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients who had undergone total knee arthroplasty surgery for the first time
* Patients who did not have a history of psychiatric problems
* Patients who were literate
* Patients who agreed to participate for the study

Exclusion Criteria:

* Patients not over 18 years
* Patients who hadn't undergone total knee arthroplasty surgery for the first time
* Patients who had a history of psychiatric problems
* Patients who weren't literate
* Patients who didn' t agree to participate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
The Quality of Life Scale Change (SF-36) | 1st day of admission to the clinic change the quality of life score at before intervention, change from baseline the quality of lıfe score at 3 days, change from baseline the quality of life score at 6 weeks
  The Quality of Life Scale (SF-36), one of the most used scales to measure quality of life; It is a self-assessment scale that can be filled in a short time and is highly sensitive.While applying the scale, individuals are asked to answer considering the last 4 weeks. The scale consists of 36 questions and 8 sub-parameters (body pain, limitation due to physical problems, limitation due to mental problems, mental well-being, fatigue, general health perception, social function and physical function). In scoring, each parameter is evaluated between 0 and 100 points. A score of 0 indicates poor health, and a score of 100 indicates good health. The higher the score, the higher the quality of life.

SECONDARY OUTCOMES:
The Function Evaluation Form Change | 1st day of admission to the clinic change the function evaluation score at before intervention, change from baseline the function evaluation score at 3 days, change from baseline the function evaluation score at 6 weeks
  The Functional Evaluation Form was developed to determine the functional status of patients who had TKA surgery and hip replacement surgery. The form consists of 8 sections and each section is scored within itself. The highest possible score is 100. The increase in score indicates the improvement in the functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Özbaş, Assist. Prof, Principal Investigator — Gazi University
Locations (1):
- Dıskapı Yıldırım Beyazıt Training and Research Hospital, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No